CLINICAL TRIAL: NCT06467123
Title: A Pilot Study Comparing Two Rehabilitation Approaches for Individuals With Irritable Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue Intervention (Experimental): Participants will attend eight sessions. During each session, participants will receive education on positions of comfort, progressing activities, and return to function. Participants will complete shoulder stretching and strengthening exercises according to a protocol.
  Interventions: Other: Tissue Intervention
- Biopsychosocial Intervention (Active Comparator): Participants will attend eight sessions. During each session, participants will receive education on pain neuroscience education, stress management, and maintaining physical activity. Participants will complete shoulder stretching and strengthening exercises according to a graded exercise protocol.
  Interventions: Other: Biopsychosocial Intervention

INTERVENTIONS:
Other: Tissue Intervention — Participants will attend eight sessions. During each session, participants will receive education on pain neuroscience education, stress management, and maintaining physical activity. Participants will complete shoulder stretching and strengthening exercises according to a graded exercise protocol.
  Arms: Tissue Intervention
Other: Biopsychosocial Intervention — Participants will attend eight sessions. During each session, participants will receive education on pain neuroscience education, stress management, and maintaining physical activity. Participants will complete shoulder stretching and strengthening exercises according to a graded exercise protocol.
  Arms: Biopsychosocial Intervention

SUMMARY:
This pilot study will assess feasibility and obtain preliminary effects of a tissue based intervention to a biopsychosocial intervention in individuals with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain intensity rated as 3/10 or higher in the past 24 hours

Exclusion Criteria:

* Non-English speaking
* Systemic medical conditions that affect sensation, such as uncontrolled diabetes
* History of shoulder surgery or fracture within the past 6 months
* blood clotting disorder, such as hemophilia
* contraindication to the application of ice ((blood pressure > 140/90 mmHg, cold urticaria, cryogobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise)
* Unable to exercise without a medical clearance (assessed on the PAR-Q+ on the first visit)
* Exceed pressure and sensory safety thresholds (assessed on the first visit)
* Categorized as low irritability (assessed on the first visit)
* currently pregnant
* currently receiving physical therapy to treat shoulder pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Report rate of adherence and adverse effects | through study completion, 4 weeks
  Number of participants who complete the study and adverse events will be reported
Report preliminary outcomes of treatment effects | through study completion, 4 weeks
  Shoulder pain intensity measured with the numeric pain rating scale will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Anderson, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided